CLINICAL TRIAL: NCT00844480
Title: Efficacy and Safety of Zoledronic Acid in Acute Spinal Cord Injury: Prevention of Bone Loss
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficulty in enrollment
Sponsor: Thomas J. Schnitzer (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Thomas J. Schnitzer, professor, Northwestern University
Organization: Northwestern University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RIC-TJS003
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Bone Loss
Keywords: spinal cord injury; osteoporosis; bone loss; zoledronic acid; bisphosphonate
MeSH Terms: conditions — Bone Diseases, Metabolic; Spinal Cord Injuries; Osteoporosis | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- zoledronic acid (Experimental)
  Interventions: Drug: zoledronic acid
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: zoledronic acid — zoledronic acid, 5mg, iv
  Other Names: Reclast, zoledronic acid
  Arms: zoledronic acid
Drug: placebo — iv
  Arms: placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled trial of zoledronic acid, 5mg, to be administered intravenously to people who have suffered an acute spinal cord fracture. The goal is to evaluate if zoledronic acid can prevent the acute bone loss seen in this population. Outcome measures will include bone density determinations over a one year period.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women
2. Age 18 years and older
3. Spinal cord injury within 8 weeks of study entry
4. ASIA AIS A or B
5. Medically stable in the opinion of their physiatrist
6. Able to have dexa performed
7. Able to return for follow-up at 6 and 12 months

Exclusion Criteria:

1. Vitamin D deficiency
2. Hypocalcemia
3. Renal insufficiency (estimated creatinine clearance <30ml/min)
4. Abnormal thyroid hormone status
5. Abnormal mental status
6. Osteoporosis at the hip or spine by dexa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-03; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Schnitzer, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Schnitzer TJ, Kim K, Marks J, Yeasted R, Simonian N, Chen D. Zoledronic Acid Treatment After Acute Spinal Cord Injury: Results of a Randomized, Placebo-Controlled Pilot Trial. PM R. 2016 Sep;8(9):833-43. doi: 10.1016/j.pmrj.2016.01.012. Epub 2016 Jan 30. PMID 26828618

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zoledronic Acid | Placebo
Started | 8 | 9
Completed | 6 | 6
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | Placebo | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (16.3) | 34.1 (15.5) | 38.9 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 5 | 8 | 13
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Bone Mass Density (BMD) at Total Hip
Description: bone mineral density measured by DXA at the total hip
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: %change in BMD from baseline
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 6 | 6
%change in BMD from baseline | -3.7 (1.0) | -12.3 (6.9)
Statistical Analysis 1: Comparison: Zoledronic Acid vs Placebo; Test type: Superiority; p = .03, t-test, 2 sided

2. Secondary Outcome: BMD at Other Skeletal Sites
Description: BMD at spine, femoral neck, distal femur, proximal tibia, heel
Time Frame: 6 months
Population: heel measurements were not performed
Measure: Mean (Standard Deviation); unit: percentage of baseline BMD
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 6 | 6
percentage of baseline BMD
  spine BMD | 2.4 (1.8) | -2.5 (2.2)
  right femoral neck BMD | -2.2 (3.4) | -8.6 (33333.5)
  distal femur | -8.2 (7.7) | -9.1 (7.1)
  proximal tibia | -3.3 (2.9) | -13.8 (10.5)
  heel: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Zoledronic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/8 | 3/9
Other Adverse Events (participants affected / at risk) | 6/8 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid (N=8) | Placebo (N=9)
baclofen pump implant (Nervous system disorders) | 0 (0) | 1 (1)
decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
infection (Infections and infestations) | 0 (0) | 1 (1) — possible urinary tract infection
hospitalization (Investigations) | 0 (0) | 1 (1) — reason for hospitalization not obtained
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid (N=8) | Placebo (N=9)
femoral fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1) | 1 (3)
fever (General disorders) | 0 (0) | 1 (2)
headache (General disorders) | 1 (1) | 1 (2)
gasric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
hypertension (Cardiac disorders) | 0 (0) | 1 (1)
chest pain (Cardiac disorders) | 1 (1) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
pressure ulcer (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
ingrown hair (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
musculoskeletall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
please see publication for discussion; small sample size major limitation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No